CLINICAL TRIAL: NCT05742997
Title: Evaluation of a Novel Diagnostic Kit for the Detection of Placental Alpha-Microglobulin-1 in the Prediction of Preterm Birth in Women Presenting With Signs and Symptoms of Preterm Labor.
Acronym: PartoSure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Principal Investigator, Caroline Van Holsbeke, Principal investigator, Ziekenhuis Oost-Limburg
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CTU202071
Record Dates: First submitted 2022-03-02; First posted 2023-02-24 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Preterm Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PartoSure (Active Comparator): Use of PartoSure to determine the risk of preterm birth
  Interventions: Device: PartoSure
- Fetal Fibronectine (fFn) (Active Comparator): Use of fFn to determine the risk of preterm birth
  Interventions: Device: Fetal Fibronectine

INTERVENTIONS:
Device: PartoSure — Diagnostic Kit for the Detection of Placental Alpha-Microglobulin-1
  Arms: PartoSure
Device: Fetal Fibronectine — Diagnostic Kit for the Detection of Fetal Fibronectine
  Arms: Fetal Fibronectine (fFn)

SUMMARY:
Currently, the American College of Obstetricians and Gynecologists (ACOG) indicate in their most recent Practice Bulletin on the Management of Preterm Labor that many tests to identify women at risk of preterm birth have been proposed and evaluated; however, only ultrasonography and fetal fibronectin testing have been shown to have benefit. Ultrasonography to determine cervical length, fetal fibronectin testing, or a combination of both may be useful in determining which women are at high risk for preterm delivery. However, their clinical usefulness may rest primarily with their ability to identify women who are least likely to deliver (i.e. their negative predictive value). Therefore, there is an urgent need for a test with a high positive predictive value in order to accurately predict imminent delivery to allow for salutary intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting for emergency obstetrical care at an emergency room or labor & delivery unit with signs, symptoms or complaints suggestive of preterm labor (PTL)

  * Uterine contractions, with or without pain
  * Intermittent lower abdominal pain
  * Dull backache
  * Pelvic pressure
  * Bleeding during the second or third trimester
  * Menstrual-like or intestinal cramping, with or without diarrhea
  * Patient is not "feeling right"
* Gestational age between 200/7 and 366/7
* Consenting to be part of the trial

Exclusion Criteria:

* Presented for regularly scheduled obstetrical care with symptoms
* < 18 years old and not emancipated consenting minor
* < 200/7 weeks of gestation or ≥ 37 weeks of gestation cervix length > 30 mm
* cervical dilatation > 3 centimeters
* overt rupture of the fetal membranes (ROM) as indicated by visualized leakage of fluid from the cervical os
* heavy vaginal bleeding
* received tocolytic medications for treatment of threatened preterm delivery prior to collection of the cervicovaginal specimens or cervical length measurements
* suspected placenta previa
* cervical cerclage in place
* a symptom not associated with idiopathic threatened preterm delivery (e.g. trauma)
* digital exam prior to specimen collection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity (SN), specificity (SP), positive predictive value (PPV) and negative predictive value | 48 hours
  Sensitivity (SN), specificity (SP), positive predictive value (PPV) and negative predictive value (NPV) for the kit for the detection of PAMG-1, cervical length measurements by trans-vaginal ultrasound (<30 mm), and contraction frequency ≥ 8 per hour.
Sensitivity (SN), specificity (SP), positive predictive value (PPV) and negative predictive value | 7 days
  Sensitivity (SN), specificity (SP), positive predictive value (PPV) and negative predictive value (NPV) for the kit for the detection of PAMG-1, cervical length measurements by trans-vaginal ultrasound (<30 mm), and contraction frequency ≥ 8 per hour.
Sensitivity (SN), specificity (SP), positive predictive value (PPV) and negative predictive value | 14 days
  Sensitivity (SN), specificity (SP), positive predictive value (PPV) and negative predictive value (NPV) for the kit for the detection of PAMG-1, cervical length measurements by trans-vaginal ultrasound (<30 mm), and contraction frequency ≥ 8 per hour.

CONTACTS AND LOCATIONS:
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No